CLINICAL TRIAL: NCT06019897
Title: Impact of Tubing Colonization on the Incidence of Central Venous Catheter Infection. Observational Study CRIC (Colonisation Des Rampes et Infection de Cathéters)
Brief Title: Impact of Tubing Colonization on the Incidence of Central Venous Catheter Infection
Acronym: CRIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202300052
Record Dates: First submitted 2023-05-25; First posted 2023-08-31 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-08

CONDITIONS: Catheter-Related Infections; Catheter Complications; Catheter Infection; Catheter-related Bloodstream Infection; Catheter Related Complication
Keywords: Catheter related infection; catheter colonization
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will swab the taps at each IV line ramp at systematic ramp changes (done every 4 days) and at catheter removal. For the multi-lumen device, swabbing is only performed upon catheter removal at the level of the one-way valves.
  After catheter removal, a flush (1 mL of 0.9% NaCl) of the midline is performed and cultured to assess for endoluminal colonization. The distal end of the CVC is sent for culture, following the usual practice of the department to monitor catheter colonization and infections. All these samples will be cultured on agar plates for microbial detection, quantification and identification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to assess the relationship between infusion system colonization (ramps or multi-lumen devices) and the occurrence of CVC infection/colonization.

This study is a prospective observational research that does not modify usual patient care. Its objective is to evaluate the relationship between infusion tubing colonization and the occurrence of central venous catheter colonization.

The only additional intervention is swabbing the taps at each IV line ramp at systematic ramp changes (done every 4 days) and at catheter removal. For the multi-lumen device, swabbing is only performed upon catheter removal at the level of the one-way valves.

After catheter removal, a flush (1 mL of 0.9% NaCl) of the midline is performed and cultured to assess for endoluminal colonization. The distal end of the CVC is sent for culture, following the usual practice of the department to monitor catheter colonization and infections.

The primary outcome measure is the proportion of colonized infusion systems based on the culture of the CVC.

The secondary objectives are to describe factors associated with CVC infections, to determine the incidence of colonization and infections in different locations of central venous catheters, to analyze the bacterial ecology based on the type of infusion system used, and to evaluate the ecological and economic impact of different devices (ramps vs. multi-lumen devices).

The secondary outcome measures are as follows:

Proportion of colonized infusion systems based on the colonization status of the CVC and the type of infusion system (ramps vs. multi-lumen devices) Proportion of colonized infusion systems based on the infection status of the CVC and the type of infusion system (ramps vs. multi-lumen devices) Duration of antibiotic treatment Weight of compounds used with each infusion system over the duration of CVC placement (ramps vs. multi-lumen devices) Calculation of material costs based on the infusion system used over the duration of CVC placement (ramps vs. multi-lumen devices)

DETAILED DESCRIPTION:
Central venous catheters (CVCs) are essential devices in the care of critically ill patients, with approximately 63% of patients admitted to intensive care being exposed to them. While they provide a safe access route for administering catecholamines or other substances unsuitable for peripheral veins, they are also associated with complications, including thrombotic and infectious events. CVC-related infections rank as the third most common nosocomial infections in the intensive care unit, representing a major public health challenge. According to the latest surveillance report on nosocomial infections in France, the incidence density is 0.61 infections per 1,000 catheter-days and 0.49 catheter-related bloodstream infections per 1,000 catheter-days. Approximately 10% of cultured catheters are found to be positive, indicating colonization. These infections are associated with an increased risk of mortality in the intensive care unit, estimated between 4% and 20%, as well as a prolonged length of stay (5-20 days) and an additional cost of approximately €10,000 per episode. Although catheter colonization has limited clinical impact, it remains a major concern due to its role as a precursor to infection. CVC infection is defined by the presence of microorganisms on the internal and/or external surface of the catheter, causing local and/or systemic infection with or without bacteremia. There are several mechanisms of infection, it is well accepted that infection begins with cutaneous colonization of the CVC, which can then spread to the intravascular part of the catheter. Another source of infection may be the colonization of infusion pathways leading to catheter colonization and infection through the "endoluminal" route. Factors associated with CVC infection include the frequency of line manipulations and the infused products. Therefore, it is recommended to minimize line manipulations, adhere to strict aseptic measures when accessing infusion lines, and regularly change (every 4 days) the infusion systems (ramps). Placing injection sites further away from the insertion site reduces the risk of contamination. The first connector tubing is never changed throughout the entire duration of CVC placement. However, there is limited data to confirm the link between infusion pathway colonization (particularly ramps used in intensive care) and catheter infection. The equipment used as infusion systems has evolved with the introduction of new devices, such as multi-lumen devices. One of these devices consists of five injection ports, each equipped with one-way valves, connected to a separate compartment in the tubing system, allowing simultaneous intravenous administration of five different active substances without mixing. This device is left in place for the entire duration of CVC placement (compared to current systems that are changed every 4 days). The objective of this study is to investigate whether there is a relationship between the colonization of infusion systems (ramps and/or multi-lumen devices) and the occurrence of CVC infection/colonization, and if this relationship varies depending on the type of device used (ramps vs. multi-lumen devices).

All adult patients hospitalized in the ICU with a CVC in place for an expected duration >2 days will be proposed to participate, in absence of oral refusal, ramps of the tubing systems will be swabed at each changes (scheduled every 4 days) and at catheter removal, in case of multi-lumen devices (edelweiss system), swabbing will be only performed upon catheter removal at the level of the one-way valves.

After catheter removal, a flush (1 mL of 0.9% NaCl) of the midline is performed and cultured to assess for endoluminal colonization. The distal end of the CVC is sent for culture, following the usual practice of the department to monitor catheter colonization and infections.

Colonization of the tubing system (ramps or multi-lumen device) will be defined as a positive culture of a swab, colonization and infection of the catheter will be defined using the CDC definitions (positiive cultutre defined as ≥10p3 CFU/ml).

Rates of catheter colonization will be compared in colonized (positive culture of a swab) or not colonized (no positiive swab culture) tubing systems. A sensibility analysis will be conducted taking into acount only the ramps and catheter colonized with the same bacterial strains.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Admitted in Surgical Intensive Care unit
* Requiring a central venous catheter for more than 48h for drug administration (central venous catheter for renal replacement therapy are excluded)

Exclusion Criteria:

* Patients < 18 years old
* Patients under legal protection
* Patients who refuse the use of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in a surgical intensive care unit and requiring a central venous catheter for drug administration
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-23 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of central venous catheter colonization according to the status colonized or not of the tubing | up to Catheter removal or up to 6 weeks
  catheter colonization is defined as a positive culture of the catheter tips ≥ 10p3 CFU/ml and compare the rates in catheter with or without a positive culture of tubiging systems

SECONDARY OUTCOMES:
Number of days without antibiotics at Day 42 (in the ICU) | up to Catheter removal or up to 6 weeks
  number of days without any antibiotic prescribed at day 42, while in the ICU. All the days outside the ICU will be considered as without antibiotics.
Incidence of colonization and infection of central venous catheter according to their site | up to Catheter removal
  we will use the CDC definition for catheter infection (with a positive culture of the catheter tips≥10p3 CFU/ml), and compare the rates in catheter with or without a positive culture of tubiging systems
Incidence of central venous catheter colonization according to the colonization of tubing and to the use or not of a multi lumen device | up to catheter removal or up to 6 weeks
  we will use the CDC definition for catheter infection (with a positive culture of the catheter tips≥10p3 CFU/ml), and compare the rates in catheter with ramps or with multilumen device
Incidence of central venous catheter infection according to the tubing colonization | up to catheter removal or up to 6 weeks
  we will use the CDC definition for catheter infection we will use the CDC definitions for catheter infection (with a positive culture of the catheter tips≥10p3 CFU/ml), and compare the rates in catheter with or without a positive culture of tubiging systems

CONTACTS AND LOCATIONS:
Overall Officials: sigismond lasocki, MD, PhD, Study Director — CHU Angers, 49033 Angers Cedex 01, France

IPD SHARING:
Plan to Share IPD: No
no plan